CLINICAL TRIAL: NCT00489021
Title: Feasibility and Outcomes of Older Patients Hospitalization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20/2007-1-HY-CTIL
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Community-Acquired Pneumonia; Exacerbation of Chronic Heart Failure; Exacerbation of Chronic Obstructive Pulmonary Disease; Cellulitis
Keywords: Subacute care; Activities of Daily Living; Cognition assessment; Mood assessment; Incontinence control
MeSH Terms: conditions — Community-Acquired Pneumonia; Cellulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: sub-acute hospitalization

SUMMARY:
Hospitalization is a traumatic event for the patient and his family at any age nevertheless in the older age. One of its consequences is the difficulty to resume previous activity of daily living especially in older (over 75 years) patients. Sub acute completes the acute phase of the hospitalization and its main purpose is to improve the patient's functional status and quality of life. There are not enough clinical trails to proof this assumption. The purpose of our study is to compare the outcome of acute and sub-acute hospitalization programs by a randomized controlled prospective intervention study. Outcome measures will comprise activity of daily living, functional status, re-hospitalization and utilization of medical services following the hospitalization.Study hypothesis is that sub-acute hospitalization will improve outcomes and will cost less.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65
* Hemodynamic, nutritional and respiratory stability
* eligibility for sub- acute hospitalization

Exclusion Criteria:

* Oncological active disease
* uncorrectable hypoxemia (oxygen saturation 90%),
* suspected myocardial ischemia
* presence of an acute illness, other than the target illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-07; Study Completion 2007-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Doron Nezer, M.D., Principal Investigator — Clalit Health Services, Israel